CLINICAL TRIAL: NCT01969552
Title: Interrelations Between FT3, FT4 and Pituitary TSH and Implications For Thyroid Hormone Treatment (IIFHT-Study)
Brief Title: Interrelations Between FT3, FT4 and Pituitary TSH
Acronym: IIFHT
Status: Completed | Type: Observational
Sponsor: Klinikum Lüdenscheid (Other)
Responsible Party: Sponsor
Other Study IDs: IIFHT-161013
Record Dates: First submitted 2013-10-16; First posted 2013-10-25 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Thyroid
Keywords: TSH, thyroid hormones, thyroid tresting, levothyroxine
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thyroid testing: Adult subjects presenting for thyroid testing or treatment

SUMMARY:
TSH plays a central role in current thyroid function testing both as a diagnostic tool and therapeutic target. Recent studies have suggested a more complex and hierarchical relationship between logTSH and FT4 over the entire functional spectrum than the widely assumed single log linear gradient (1-4). Our group has also shown a disjoint between pituitary TSH and FT3 serum levels being operative under conditions of levothyroxine monotherapy (5).

The present prospective observational study aims at confirming some of these findings and exploring additional factors other than TSH that may be important in shaping the interrelation of thyroid parameters and modulating thyroidal activity in health and disease.

To this purpose, unselected patients presenting for thyroid testing or treatment to a specialised unit at a teaching hospital will be prospectively studied to assess the interplay of FT3, FT4 and TSH under various conditions, and to evaluate various thyroidal and non-thyroidal influences, such as disease entity, thyroid volume, deiodinase activity, thyroid medication, surgery, radioiodine treatment, age, BMI, smoking on pituitary set-point and homeostatic equilibria.

DETAILED DESCRIPTION:
Study Design: Prospective observational cross-sectional monocentre study

Eligible Patients: Adult subjects presenting for thyroid testing or treatment to the Department of Nuclear Medicine, Klinikum Luedenscheid, Luedenscheid, Germany.

Inclusion criteria: All consecutively seen subjects who consent to precipitate and to fill out a questionnaire, which represent the full functional spectrum, as seen in a praxis setting.

Exclusion criteria from analysis: Missing consent, severe illness that may be associated with euthyroid sick syndrome (non-thyroidal illness syndrome), pregnancy, pituitary and hypothalamic disorders as well as medication that may impair pituitary thyroid hormone feedback

Methods: Except for a detailed questionnaire the study includes routine work-up, established standard procedures for diagnosis and standard care for treatment of thyroid disease Patient history and physical examination Detailed questionnaire on disease history and medication Measurement of thyroid function parameters and autoantibodies Ultrasound of thyroid gland and scintigraphy where required

Statistical analysis includes group comparisons, correlations, generalised linear models with multiple covariates and more advanced modelling techniques of feedback control and FT3- FT4-TSH interrelations, as previously described (4, 5, 6).

Outcome Measures: Group comparisons among treated patients and untreated subjects and various disease entities, modelling of lnTSH interactions with FT4 and FT3,influence of clinically relevant covariates on FT3-FT4-TSH interrelations and equilibria.

Estimated Enrolment : approx. 1500 patients

Estimated Duration: approx. 12 months

Ethical approval: Ethical Committee of the University of Muenster, Muenster, Germany

Sponsor: none

Financial Support: none

Conflicts of Interest: none

ELIGIBILITY:
Inclusion Criteria:

* All consecutively seen subjects who consent to precipitate and to fill out a questionnaire, which represent the full functional spectrum, as seen in a praxis setting.

Exclusion Criteria:

* Missing consent, severe illness that may be associated with euthyroid sick syndrome (non-thyroidal illness syndrome), pregnancy, pituitary and hypothalamic disorders as well as medication that may impair pituitary thyroid hormone feedback.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects presenting for thyroid testing or treatment to the Department of Nuclear Medicine, Klinikum Luedenscheid, Luedenscheid, Germany.
Sampling Method: Probability Sample
Enrollment: 1912 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pituitary setpoint and thyroid hormone equilibria | Baseline
  According to our previous work, the states of hypothyroidism, euthyroidism and hyperthyroidism can be regarded as differently regulated entities. The present study assesses modulators that influence pituitary thyroid feedback control and impact on the pituitary setpoint and hormonal equilibria. The measure is change in circulating levels of TSH (mU/L) per change in FT4 (nmol/L) or FT3 (pmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Larisch, Prof, Principal Investigator — Klinikum Lüdenscheid Department of Nuclear Medicine; Rudolf Hoermann, Prof, Study Chair — Klinikum Luedenscheid Department of Nuclear Medicine
Locations (1):
- Department of Nuclear Medicine Klinikum Luedenscheid, Lüdenscheid, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Hoermann R, Eckl W, Hoermann C, Larisch R. Complex relationship between free thyroxine and TSH in the regulation of thyroid function. Eur J Endocrinol. 2010 Jun;162(6):1123-9. doi: 10.1530/EJE-10-0106. Epub 2010 Mar 18. PMID 20299491
- [Background] Midgley JE, Hoermann R, Larisch R, Dietrich JW. Physiological states and functional relation between thyrotropin and free thyroxine in thyroid health and disease: in vivo and in silico data suggest a hierarchical model. J Clin Pathol. 2013 Apr;66(4):335-42. doi: 10.1136/jclinpath-2012-201213. Epub 2013 Feb 19. PMID 23423518
- [Background] Clark PM, Holder RL, Haque SM, Hobbs FD, Roberts LM, Franklyn JA. The relationship between serum TSH and free T4 in older people. Postgrad Med J. 2012 Nov;88(1045):668-70. doi: 10.1136/postgradmedj-2011-200433rep. PMID 23097057
- [Background] Hadlow NC, Rothacker KM, Wardrop R, Brown SJ, Lim EM, Walsh JP. The relationship between TSH and free T(4) in a large population is complex and nonlinear and differs by age and sex. J Clin Endocrinol Metab. 2013 Jul;98(7):2936-43. doi: 10.1210/jc.2012-4223. Epub 2013 May 13. PMID 23671314
- [Background] Hoermann R, Midgley JE, Larisch R, Dietrich JW. Is pituitary TSH an adequate measure of thyroid hormone-controlled homoeostasis during thyroxine treatment? Eur J Endocrinol. 2013 Jan 17;168(2):271-80. doi: 10.1530/EJE-12-0819. Print 2013 Feb. PMID 23184912
- [Background] Dietrich JW, Landgrafe G, Fotiadou EH. TSH and Thyrotropic Agonists: Key Actors in Thyroid Homeostasis. J Thyroid Res. 2012;2012:351864. doi: 10.1155/2012/351864. Epub 2012 Dec 30. PMID 23365787